CLINICAL TRIAL: NCT04314128
Title: Assessment of Raised Intracranial Pressure in Patients With Idiopathic Intracranial Hypertension by Optic Nerve Sheath Diameter and Transcranial Doppler Measurements
Brief Title: Assessment of ICP in Idiopathic Intracranial Hypertension Using Transocular Ultrasound and Transcranial Doppler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Johanne Severinsen, Medical Doctor, Danish Headache Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-19029542
Record Dates: First submitted 2020-03-12; First posted 2020-03-19 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Idiopathic Intracranial Hypertension
MeSH Terms: conditions — Pseudotumor Cerebri | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Intervention Model Description: Single group, prospective cohort study with healthy controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients suspected of IIH at baseline (Other): Intervention: TOS and TCD measurements at baseline, and at routine follow-ups.
  Healthy controls will be recruited to match the patients.
  Interventions: Diagnostic Test: TOS and TCD

INTERVENTIONS:
Diagnostic Test: TOS and TCD — TOS: Transorbital sonography TCD: Transcranial Doppler

SUMMARY:
Idiopathic Intracranial Hypertension (IIH) is a rare disease, primarily affecting overweight females of child-bearing age. Patients suffer from increased intracranial pressure (ICP), typically resulting in headaches, visual disturbances and bilateral papilledema, pulsatile tinnitus and cognitive deficits. The disease is difficult to diagnose, treat and monitor. The only current method of measuring the ICP in day-to-day clinical practice is by lumbar puncture. This procedure is invasive, and often painful for the patient. There is an unmet need of methods that can reliable measure or estimate ICP in a non-invasive manner. Ultrasound is one such potential method, and the aim of this study is to investigate the use of ocular ultrasound and transcranial doppler to measure or estimate ICP.

DETAILED DESCRIPTION:
This study is a prospective cohort study. Investigators plan to include 50 patients in whom the IIH-diagnosis is suspected. Patients are referred from general practitioners, neurologists or ophthalmologists to the Danish Headache Center or admitted to the Neurology ward when the IIH diagnosis is suspected.

As part of an established routine clinical work-up to establish the diagnosis of IIH, all patients will undergo (according to the Friedman criteria) the following examinations:

A)

1. An interview (history taking) and clinical examination
2. Routine laboratory tests (blood tests)
3. Ophthalmological examination
4. Lumbar puncture with measurement of the ICP
5. Magnetic resonance imaging (MRI) of the brain

Additionally the following investigations will be performed at baseline (before and after lumbar puncture):

B) Transorbital sonography (TOS) C) Transcranial Doppler When the patient is seen at the clinic for their regular follow-up visits the same measurements will be done.

A control group of healthy participants (NR=25) will be included in whom TOS (B) and TCD (C) will be performed in order to compare the values between the patient group (IIH) and control group. Controls will be included to match the patients according to BMI, age and gender.

All ultrasound images- and films will be saved, and evaluated by a blinded investigator.

ELIGIBILITY:
PATIENT GROUP (ARM 1):

Inclusion Criteria:

* Age 18-65
* Patients in whom the IIH diagnosis is suspected/or confirmed
* The diagnosis of migraine with or without aura or tension-type headache is allowed as a comorbid headache type.
* Participants must read and understand the Danish language, or have an official interpreter present to be able to understand the work-up and sign the participation consent for the study

Exclusion Criteria:

* Pregnant or breastfeeding females
* Patients who do not need a diagnostic lumbar puncture at the time of evaluation
* Patients treated with acetazolamide, topiramate or furosemide for IIH or suspected IIH before inclusion in the study (baseline)
* Any other primary or secondary headache diagnosis than migraine with or without aura or tension type headache as a comorbid disorder
* Patients in whom the examination cannot be performed due to anatomical reasons such as severe head dysmorphia or severe ophthalmological diseases
* Participants with secondary causes of raised intracranial pressure, or patients that have been treated for such (e.g. brain tumor, hydrocephalus, stroke or severe head injury)
* Participants with known atherosclerotic disease or known heart disease

CONTROL GROUP (ARM 2):

Inclusion criteria:

* Age 18-65
* Healthy persons who do not suffer from any form of primary headache except infrequent tension-type headache
* Participants must read and understand the Danish language or have an official interpreter present to be able to sign the participation consent for the study.

Exclusion criteria:

* Pregnant or breastfeeding females
* Participants in whom the examination cannot be performed due to anatomical reasons such as severe head dysmorphia or severe ophthalmological diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Correlation between opening pressure and ONSD | 1 year
  Optic nerve sheath diameter (ONSD) potential correlation with opening pressure.
Correlaton between opening pressure and ONSD/ETD ratio | 1 year
  ONSD/ETD (external transverse diameter) ratio and potential correlation with opening pressure.
Comparison of ONSD in IIH and healthy controls | 1 year
  Comparison of ONSD in patients with elevated ICP (IIH) and healthy controls, age- sex and BMI matched.

SECONDARY OUTCOMES:
Optic disc elevation | 1 year
  Optic disc elevation measured by ultrasound in IIH compared with healthy controls
ONSD diameter on MR c in patients with IIH | 1 year
  ONSD and correlation with ONSD on orbital MRI.
Changes in the optic nerve (ONSD) | 1 month
  Changes in ONSD after 1 month
Changes in the optic nerve (ONSD) | 6 months
  Changes in ONSD after 6 months
Changes in the optic nerve (ODE) | 1 month
  Changes in ODE (optic disc elevation) after 1 month
Changes in the optic nerve (ODE) | 6 months
  Changes in ODE(optic disc elevation) after 6 months
TCD (PI - pulsatility index) in patients with IIH | 2 years
  Evaluation of pulsatility index for major intracranial arteries (PI) using doppler ultrasound in patients with raised intracranial pressure (IIH) compared with normal values.
TCD (MBFV - mean blood flow velocity) in patients with IIH | 2 years
  Evaluation of mean blood flow velocity (MBFV) for major intracranial arteries using doppler ultrasound in patients with raised intracranial pressure (IIH) compared with normal values.
TCD (RI - resistance index) in patients with IIH | 2 years
  Evaluation of resistance index (RI) for major intracranial arteries using doppler ultrasound in patients with raised intracranial pressure (IIH) compared with normal values.
Neuro-ophthalmological evaluation of papilledema versus ultrasound evaluation of the optic nerve | 2 years
  Papilledema and the optic nerve is usually evaluated by neuro-ophthalmologists in patients with IIH. Investigators will compare this evaluation with the assessment made by TOS ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Rigmor Jensen, Dr.med., Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No